CLINICAL TRIAL: NCT00766883
Title: A Phase II Clinical Trial to Determine the Effectiveness of Problem Solving Education in Caregivers and Patients During Allogeneic HSCT
Brief Title: Problem-Solving Education for Caregivers and Patients During Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080220; 08-CC-0220
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2017-09-28

CONDITIONS: Distress; Hematopoietic Stem Cell Transplantation
Keywords: Allogeneic HSCT; Psychosocial Distress; Coping; Cognitive Behavior Therapy; Self Efficacy; Allogeneic Stem Cell Transplant

INTERVENTIONS:
Behavioral: Problem Solving Education

SUMMARY:
This study will examine the effectiveness of problem-solving education for patients who are undergoing a stem cell transplant and their caregivers. The emotional stress of transplant extends beyond patients to their caregivers; this study will identify the type of education that will be most helpful to transplant caregivers.

Adult patients undergoing stem cell transplant at the NIH s Clinical Center and their adult caregivers are eligible for this study. The caregiver must be caring for the patient from before hospital admission for the procedure until 6 weeks following the transplant. Both patient and caregiver must be able to read and speak English.

Patients and caregivers have three education sessions (in addition to the routine transplant education provided at the Clinical Center) and complete three study questionnaires as follows:

* Questionnaires: The questionnaires vary somewhat for patient and caregiver, but include information on demographics (e.g., sex, race, marital status, education level), distress, lifestyle, relationship with the caregiver/patient, confidence level, symptoms, pain, fatigue and sleep quality. Questionnaires are completed before the patient undergoes the transplant (and before attending any education sessions), before the patient is discharged from the hospital and 6 weeks after hospital discharge.
* Education sessions: The 60-minute sessions are designed to teach problem-solving strategies by looking at problems in a new way and learning effective communication skills. The sessions are conducted before the patient is discharged from the hospital, 1 week after discharge and 3 weeks after discharge.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (HSCT) generates multiple symptoms and problems that can vary in complexity. Although it seems evident that patients and caregivers experience clinically significant levels of psychological distress, few intervention studies have been explored to address this concern in this population.

Problem-solving is an essential skill for individuals to successfully cope. Increased problem-solving skill has been shown to decrease psychological distress and may improve symptom distress and health related quality of life (QOL). The COPE (Creativity, Optimism, Planning, and Expert Information) problem-solving education (PSE) intervention has demonstrated benefit and has been reported as a positive therapy by cancer patients and their families. Only one study has reported the application of this intervention in the acute care setting and our previous pilot study has been the only one done with patients and caregivers undergoing allogeneic HSCT.

Based on the findings from our pilot study and recent published reports, this study is designed to determine preliminary efficacy of problem solving education by increasing self-efficacy in caregivers during allogeneic HSCT. In addition, this study will explore factors associated with change in caregiver self-efficacy and distress such as demographics, clinical variables, mutuality, caregiver reaction, sleep quality, fatigue and health behaviors.

This is a phase two clinical trial applying a prospective repeated measure design. Subjects will be accrued to this protocol if they agree to participation in an allogeneic HSCT at the Clinical Center, NIH, are greater than 18 years old, able to read English and able to comprehend the investigational nature of the study. Patient volunteers must have at least one caregiver throughout the study period. A sample of at least 71 caregivers is needed to adequately evaluate the effectiveness of the PSE intervention. In order to achieve a sample of 71 caregivers 50 transplant patients will be recruited.

Each caregiver (and patient) will be scheduled for three individualized PSE intervention sessions (study intervention) in addition to the usual care group education. Three surveys will be administered to all study participants. The baseline questionnaires will be administered twice; once prior to allogeneic HSCT and again directly before the first PSE, at the time of initial discharge from the hospital. The post-intervention questionnaires will be administered 6 weeks post discharge. There will be no long term follow-up after the intervention period. Questionnaires include: Distress Thermometer, Family Caregiving Inventory Mutuality Scale, Health-Promoting Lifestyle Profile II, Cancer Self-Efficacy scale, Brief Symptom Inventory, Caregiver Reaction Assessment, Pittsburgh Sleep Quality Index and the Multidimensional Fatigue Symptom Inventory-Short Form. In addition, the subjects will participate in a semi-structured interview at the end of the study and the interventionist will complete a log that tracks subject attendance, session length, and discrepancy between planned and actual session date and time. Quantitative and qualitative analysis techniques will be used in this study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients:

* Receiving their first allogeneic HSCT at the CC, NIH.
* Age greater than or equal to 18 years old.
* Ability to comprehend the investigational nature of the study and provide informed consent.
* Able to read and speak English.
* Adult caregiver(s) available and/or living with transplant recipient.
* Caregiver(s) agrees to participate in the study.

Caregiver(s):

* Age greater than or equal to 18 years old.
* Ability to comprehend the investigational nature of the study and provide informed consent.
* Able to read and speak English.
* Agrees to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2008-09-29; Primary Completion 2010-12-15 (Actual); Study Completion 2010-12-15 (Actual)

PRIMARY OUTCOMES:
To determine the effect of a PSE intervention on self-efficacy (a sense of control of oneself) in caregivers during the experience of an allogeneic HSCT.

SECONDARY OUTCOMES:
To determine the effect of a PSE intervention on self-efficacy (a sense of control of oneself) in patients during the experience of an allogeneic HSCT.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret F Bevans, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Goldman JM, Horowitz MM. The international bone marrow transplant registry. Int J Hematol. 2002 Aug;76 Suppl 1:393-7. doi: 10.1007/BF03165291. PMID 12430889
- [Background] Tabbara IA, Zimmerman K, Morgan C, Nahleh Z. Allogeneic hematopoietic stem cell transplantation: complications and results. Arch Intern Med. 2002 Jul 22;162(14):1558-66. doi: 10.1001/archinte.162.14.1558. PMID 12123398
- [Background] Thomas ED, Blume KG. Historical markers in the development of allogeneic hematopoietic cell transplantation. Biol Blood Marrow Transplant. 1999;5(6):341-6. doi: 10.1016/s1083-8791(99)70010-8. No abstract available. PMID 10595811
- [Derived] Sundaramurthi T, Wehrlen L, Friedman E, Thomas S, Bevans M. Hematopoietic Stem Cell Transplantation Recipient and Caregiver Factors Affecting Length of Stay and Readmission. Oncol Nurs Forum. 2017 Sep 1;44(5):571-579. doi: 10.1188/17.ONF.571-579. PMID 28820507